CLINICAL TRIAL: NCT02362633
Title: Effect of Long-term Transcranial Direct Current Stimulation (tDCS) on Appetite Control Related Brain Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungbuk National University (Other)
Responsible Party: Principal Investigator, Hyung Jin Choi, Clinical Assistant Professor, Chungbuk National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-07-018
Record Dates: First submitted 2015-02-02; First posted 2015-02-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Real tDCS (Experimental): Subjects will receive real tDCS treatment for ten times for two weeks (five times per week).
  Interventions: Device: real tDCS
- Sham tDCS (Sham Comparator): Subjects will receive sham tDCS treatment for ten times for two weeks (five times per week).
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: real tDCS — For active tDCS, a 2 mA current will be delivered for 20 minutes with 20 second up and down ramp times. The anodal electrode will be placed on the right DLPFC (F4; 10-20 EEG system), and the cathode electrode will be placed on the left DLPFC (F4;10-20 EEG system), which is known to be related to cognitive function. The electrodes used for tDCS are saline-soaked sponges (25 cm2).
  Arms: Real tDCS
Device: sham tDCS — Sham tDCS will be delivered for 20 minutes. The anodal electrode will be placed on the right DLPFC (F4; 10-20 EEG system), and the cathode electrode will be placed on the left DLPFC (F4;10-20 EEG system), which is known to be related to cognitive function. The electrodes used for tDCS are saline-soaked sponges (25 cm2).
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to investigate the long-term effect of Transcranial Direct Current Stimulation (tDCS) on appetite control related brain regions.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is emerging tool for brain modulation in a variety of clinical conditions. In addition, recent neuroimaging studies suggest that modifying the activity of brain circuits involved in eating behavior could provide therapeutic benefits in obesity.

The investigators aim to assess whether long-term modulation of the dorsolateral prefrontal cortex (DLFPC) using tDCS, modifies behavioral response and brain activity while watching visually presented food cues and taste cues in obese subjects.

Subjects will be randomly divided into sham and real tDCS arms. Subjects will receive sham or real tDCS ten times. Subjects will be investigated before and after sham or real tDCS interventions. Subjects will perform functional MRI experiments with visual and taste food cues. Questionnaire with behavior measures, body compositions, blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 26 kg/m2

Exclusion Criteria:

* History of brain trauma, epilepsy, or other neurological problems

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Regional brain activity measured by blood-oxygen-level dependent (BOLD) signal of functional MRI | Day 14 (After ten interventions)
  3T MR scanner with Echo Planar Imaging(EPI) capability(Magnetom, Siemens Medical System)

SECONDARY OUTCOMES:
Behavior outcomes on the visual analog scale | Day 14 (After ten interventions)
  Hunger related visual analogue scale (VAS) - 8 items (Flint et al., 2000) Mood related visual analogue scale (VAS) - 16 items (Fregni et al., 2008)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University, Cheongju-si, North Chungcheong, South Korea